CLINICAL TRIAL: NCT06749756
Title: Study on the Improvement of Microcirculation in Patients With Sepsis by Vitamin B6, Vitamin B12 and Vitamin C
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fan Zeng (Other)
Responsible Party: Sponsor-Investigator, Fan Zeng, Deputy chief physician, Sichuan Cancer Hospital and Research Institute
Organization: Sichuan Cancer Hospital and Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: No. 742-1in2024ofLunShen(Yan）
Record Dates: First submitted 2024-12-07; First posted 2024-12-27 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Ascorbic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental group (Experimental): In addition to the basic treatment of sepsis, intravenous injection of vitamin B6 300mg qd Vitamin B12 0.5mg q6h, vitamin C 50mg/kg q6h for 4 days.
  Interventions: Drug: vitamin B6+ Vitamin B12 +vitamin C
- Control group 1 (Active Comparator): In addition to the basic treatment of sepsis, vitamin B6 300mg qd and vitamin B12 0.5mg q6h were given intravenously for 4 days.
  Interventions: Drug: vitamin B6+ Vitamin B12
- Control group 2 (Active Comparator): On the basis of the basic treatment of sepsis, intravenous vitamin C 50mg/kg q6h was given for 4 days.
  Interventions: Drug: vitamin C
- Control group 3 (Active Comparator): The same dose of placebo (0.9% sodium chloride solution) was administered on top of the sepsis base treatment for 4 days.
  Interventions: Drug: 0.9%Nacl

INTERVENTIONS:
Drug: vitamin B6+ Vitamin B12 +vitamin C — In addition to the basic treatment of sepsis, intravenous injection of vitamin B6 300mg qd Vitamin B12 0.5mg q6h, vitamin C 50mg/kg q6h for 4 days.
  Arms: Experimental group
Drug: vitamin B6+ Vitamin B12 — In addition to the basic treatment of sepsis, vitamin B6 300mg qd and vitamin B12 0.5mg q6h were given intravenously for 4 days.
  Arms: Control group 1
Drug: vitamin C — On the basis of the basic treatment of sepsis, intravenous vitamin C 50mg/kg q6h was given for 4 days.
  Arms: Control group 2
Drug: 0.9%Nacl — The same dose of placebo (0.9% sodium chloride solution) was administered on top of the sepsis base treatment for 4 days.
  Arms: Control group 3

SUMMARY:
Sepsis is a kind of disease with high morbidity and mortality in ICU. At present, there is no specific treatment, and its pathogenesis is mainly excessive oxidative stress. Anti-inflammatory, antioxidant and immune-regulating drugs may produce better therapeutic effects, while vitamin B6, vitamin B12 and vitamin C have anti-inflammatory, antioxidant and immune-regulating effects. The purpose of this study was to investigate whether vitamin B6, vitamin B12 combined with vitamin C can improve the microcirculation and organ dysfunction in patients with sepsis, and improve the survival rate of patients with sepsis. The study included 296 patients who met the inclusion criteria. After randomization, the experimental group was given intravenous vitamin B6 300mg qd in addition to the basic treatment of sepsis Vitamin B12 0.5mg q6h, vitamin C 50mg/kg q6h for 4 days. Control group 1 was given vitamin B6 300mg qd and vitamin B12 0.5mg q6h intravenously for 4 days. Control group 2 was injected with vitamin C 50mg/kg q6h intravenously for 4 days. Control group 3: The same dose of placebo (0.9% sodium chloride solution) was administered for 4 days. After medication, sublingual microcirculation image and radial artery resistance index of snus pit were detected and recorded according to the time required by the study protocol. The duration of use of pressor drugs, ventilator days, ICU stay, 28-day mortality, capillary refill time, changes in SOFA score and APACHEII score on day 3 and day 7 compared with baseline values at randomization, daily veno-arterial carbon dioxide differential pressure (GAP) and central venous oxygen saturation were recorded. After the end of the experiment, statistical analysis of the data was carried out to further explore the test results

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and < 85 years old
2. Admitted to ICU
3. Diagnosis of patients with SEPSIS 3.0 (diagnostic criteria) 4, SOFA score is 2-13 points

5. Obtain the informed consent of the subject or his family

Exclusion Criteria:

1. Patients have absolute contraindications such as vitamin allergy
2. Patients with a history of gout
3. Death is expected within 24 hours
4. Pregnant women
5. Use hydroprednisone or other equivalent dose hormones > 200mg/d within 24 hours
6. Without the informed consent of the patient or his/her representative
7. Patients with a history of scleroderma
8. Patients with a history of vasculitis
9. Patients with oral mucosal diseases
10. Patients with severe difficulty in opening their mouth and unable to detect sublingual microcirculation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Estimated)
Dates: Start 2025-02-10 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Improvement of microcirculation | At 0 hour, 6hours, 24hours, 48hours, 4 days, and 7 days after initiation of administration.
  Sublingual microcirculation index (including perfusion vessel density (PVD) and total vessel density (TVD)) was measured after initiation of administration.
Improvement of microcirculation | At 0 hour, 6hours, 24hours, 48hours, 4 days, and 7 days after initiation of administration.
  The radial artery resistance index of snus pit was measured after the start of administration.

SECONDARY OUTCOMES:
The duration of the patient's use of pressor drugs | 4 days
  Duration of pressor drug use during the patient's trial medication
Number of days on ventilator | 28 days
  The number of days the patient was ventilator-ventilated within 28 days
ICU stay | 28 days
  Patient's 28-day ICU stay
28-day mortality | 28 days
  28-day mortality
Capillary refill time | 4 days
  Capillary refill time during trial medication
Changes in SOFA score | 7 days
  Changes in SOFA scores on day 3 and day 7 compared with baseline values at randomization.The SOFA Score (Sequential Organ Failure Assessment Score) is a scoring system used to assess the severity of organ dysfunction in critically ill patients. It consists of six systems: respiratory, blood, liver, cardiovascular, nervous and kidney, with each system scored according to the degree of dysfunction on a scale of 0 (normal) to 4 (severe impairment or failure). The score of SOFA is closely related to the mortality and prognosis of patients. The higher the score, the higher the mortality.
Changes in APACHEII score | 7 days
  Changes in APACHEII scores on day 3 and day 7 compared with baseline values at randomization.The Apache II score, also known as the Acute Physiological and Chronic Health Assessment (APACHE II), is a scoring system used to assess the severity of a critically ill patient's condition and predict prognosis. The theoretical maximum value is 71 points, and the higher the score, the more severe the disease, the worse the prognosis and the higher the fatality rate.
Daily change of veno-arterial carbon dioxide differential pressure (GAP) | 4 days
  Daily change of veno-arterial carbon dioxide differential pressure (GAP)
Daily change of central venous oxygen saturation (Scv02) | 4 days
  Daily change of central venous oxygen saturation (Scv02)

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wald EL, Badke CM, Hintz LK, Spewak M, Sanchez-Pinto LN. Vitamin therapy in sepsis. Pediatr Res. 2022 Jan;91(2):328-336. doi: 10.1038/s41390-021-01673-6. Epub 2021 Jul 31. PMID 34333556
- [Result] Giustina AD, Danielski LG, Novochadlo MM, Goldim MPS, Joaquim L, Metzker KLL, Carli RJ, Denicol T, Cidreira T, Vieira T, Petronilho F. Vitamin B6 reduces oxidative stress in lungs and liver in experimental sepsis. An Acad Bras Cienc. 2019 Dec 2;91(4):e20190434. doi: 10.1590/0001-3765201920190434. eCollection 2019. PMID 31800708
- [Result] Wang Y, Lu WL, Feng WM, Xu W, Liu LH, He LM. RENAL PROTECTIVE EFFECT AND CLINICAL ANALYSIS OF VITAMIN B 6 IN PATIENTS WITH SEPSIS. Shock. 2024 Jun 1;61(6):841-847. doi: 10.1097/SHK.0000000000002329. Epub 2024 Apr 26. PMID 38691102
- [Result] Zhao W, Zhang J, Lu Y, Wang R. The vasorelaxant effect of H(2)S as a novel endogenous gaseous K(ATP) channel opener. EMBO J. 2001 Nov 1;20(21):6008-16. doi: 10.1093/emboj/20.21.6008. PMID 11689441
- [Result] Patel JJ, Willoughby R, Peterson J, Carver T, Zelten J, Markiewicz A, Spiegelhoff K, Hipp LA, Canales B, Szabo A, Heyland DK, Stoppe C, Zielonka J, Freed JK. High-Dose IV Hydroxocobalamin (Vitamin B12) in Septic Shock: A Double-Blind, Allocation-Concealed, Placebo-Controlled Single-Center Pilot Randomized Controlled Trial (The Intravenous Hydroxocobalamin in Septic Shock Trial). Chest. 2023 Feb;163(2):303-312. doi: 10.1016/j.chest.2022.09.021. Epub 2022 Sep 26. PMID 36174744
- [Result] Fisher BJ, Seropian IM, Kraskauskas D, Thakkar JN, Voelkel NF, Fowler AA 3rd, Natarajan R. Ascorbic acid attenuates lipopolysaccharide-induced acute lung injury. Crit Care Med. 2011 Jun;39(6):1454-60. doi: 10.1097/CCM.0b013e3182120cb8. PMID 21358394
- [Result] Sevransky JE, Rothman RE, Hager DN, Bernard GR, Brown SM, Buchman TG, Busse LW, Coopersmith CM, DeWilde C, Ely EW, Eyzaguirre LM, Fowler AA, Gaieski DF, Gong MN, Hall A, Hinson JS, Hooper MH, Kelen GD, Khan A, Levine MA, Lewis RJ, Lindsell CJ, Marlin JS, McGlothlin A, Moore BL, Nugent KL, Nwosu S, Polito CC, Rice TW, Ricketts EP, Rudolph CC, Sanfilippo F, Viele K, Martin GS, Wright DW; VICTAS Investigators. Effect of Vitamin C, Thiamine, and Hydrocortisone on Ventilator- and Vasopressor-Free Days in Patients With Sepsis: The VICTAS Randomized Clinical Trial. JAMA. 2021 Feb 23;325(8):742-750. doi: 10.1001/jama.2020.24505. PMID 33620405